Title

Advanced Directives in Palliative Care: physician's role on caregiver's

empowerment as patient's surrogates.

Date: 18th April 2018

## Informed Consent to Participate in Research (Patient - A)

| DAVPAL Number | A |
|---------------|---|
|---------------|---|

Please read the following information carefully. If you think something is incorrect, or unclear, don't hesitate to ask for more information. If you agree with the proposal made to you, please sign this document.

**Title**: DAVPAL Study (Advanced Directives in Palliative Care)

**Context**: Research study for the elaboration of a Doctoral Thesis in Palliative Care on the Faculty of Medicine of the University of Porto, under the supervision of Professor Rui Nunes.

Researcher: Catarina Sampaio Martins

Medicine Doctor in Anesthesiology and Palliative Care

**Description of the Study**: The DAVPAL Study is a prospective, randomized, controlled, patient-blind study, involving patients referred to the Palliative Care consultation at the Hospital Center of Tràs-os-Montes and Alto Douro, and their families, whose main objective is to assess the ability of the palliative physician to improve the concordance between patients and their family members, regarding the patients' Advance Directives.

The patients will be asked to:

- ✓ Appoint a "health surrogate" (who also consents to participate in the study)
- ✓ Complete socio-demographic variable questionnaires
- ✓ Fill in the official Advance Directives template
- ✓ Complete questionnaires validated for the Portuguese population
- ✓ Undergone an interview with the Palliative doctor

**Conditions**: The DAVPAL Study is financed exclusively by the researcher, with no payment or compensation from the interveners. Participation in the DAVPAL study is voluntary, with no prejudice or other harm for patients who refuse to participate. The DAVPAL study was approved by the Ethics Committee of the Centro Hospitalar of Tràs-os-Montes and Alto Douro.

**Confidentiality and Anonymity**: Data collected in the DAVPAL Study will be confidential, anonymous, and used exclusively for the present study.

Thank you for your cooperation.

## Catarina Sampaio Martins

Medicine Doctor in Anesthesiology and Palliative Care on Centro Hospitalar of Tràs-os-Montes and Alto Douro

Email: <u>catarinasamp@gmail.com</u> Phone number: 925484026

| Researcher Signature: |
|-----------------------|
| • |

<u>catarinasamp@gmail.com</u> Phone number: 925484026

## I declare that:

- ✓ I have read and understood this document, as well as the verbal information provided to me by the researcher;
- ✓ I understood the explanation given to me about the research that is intended to be carried out, as well as the study in which I will be included;
- ✓ I had the opportunity to ask all the questions I thought necessary, having received a satisfactory answer;
- ✓ I understood that I have the right to refuse participation in the study at any time, without the need to give any explanation and without this having the effect of causing any harm to the assistance provided to me.

Thus, I accept to participate in this study, and I allow the use of the data that I voluntarily provide, trusting that it will only be used for this investigation, and in the guarantees of confidentiality and anonymity given to me by the researcher.

| Patient Name: |
|--------------------------------------------------|
| Signature: |
| Date:/ |
| If other than the patient: |
| Name: |
| Identification card numberValidity: |
| Parentage or affinity to the patient |
| Signature |
| Date:/ |
| Researcher Signature: (CATARINA SAMPAIO MARTINS) |
| Profissional Number: 39138 |
| Date:/ |

This document consists of 2 pages and is done in duplicate: One way for the Investigator, another for the person who consents.